CLINICAL TRIAL: NCT01726582
Title: A Prospective Phase II Trial of Molecular Profiling to Guide Neoadjuvant Therapy for Resectable and Borderline Resectable Adenocarcinoma of the Pancreas
Brief Title: Pancreas Cancer: Molecular Profiling as a Guide to Therapy Before and After Surgery ("Personalized Medicine")
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Susan Tsai, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCW 15565; Advancing a Healthier WI (Other Grant/Funding Number: Medical College of Wisconsin FP180 AHW Endowment); FP 7718 (Other Grant/Funding Number: Froedtert Hospital Foundation)
Record Dates: First submitted 2011-12-28; First posted 2012-11-15 (Estimated); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: pancreas; adenocarcinoma; molecular profile; molecular profiling; pancreatic cancer; pancreas cancer; cancer; molecular target; pancreas head; pancreas neck; pancreas uncinate; pancreas body; pancreas tail
MeSH Terms: conditions — Adenocarcinoma; Pancreatic Neoplasms; Neoplasms | interventions — folfirinox; IFL protocol; Gemcitabine; Irinotecan; gemcitabine-oxaliplatin regimen; Cisplatin; Capecitabine; 130-nm albumin-bound paclitaxel; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Milestones related to therapy (Experimental): Milestone 1: Targeted chemotherapy prior to surgery: 8 weeks targeted chemotherapy; restaging.
  Milestone 2: Before surgery: Chemoradiotherapy (cRXT); restaging Milestone 3: Before surgery: 8 weeks targeted chemotherapy; restaging; chemoradiotherapy (cXRT); restaging.
  Milestone 4: standard FOLFIRINOX chemotherapy prior to surgery: 8 weeks FOLFIRINOX (standard chemotherapy); restaging; standard chemoradiotherapy (cXRT); restaging.
  Milestone 5: After surgery: 8 weeks targeted chemotherapy; restaging; chemoradiotherapy (cXRT); restaging.
  Milestone 6: Gemcitabine after surgery: 8 weeks standard Gemcitabine (chemotherapy); restaging; chemoradiotherapy (cXRT); restaging.
  Milestone 7: After surgery: chemoradiotherapy (cXRT); restaging. Milestone 8: Gemcitabine after surgery: 8 weeks Gemcitabine (chemotherapy); restaging; 8 weeks Gemcitabine (chemotherapy); restaging.
  Milestone 9: No additional therapy after surgery. Milestone 10: After surgery no additional treatment.
  Interventions: Drug: Milestone 1: Targeted chemotherapy prior to surgery; Radiation: Milestone 2: Chemoradiotherapy (cXRT); Drug: Milestone 3: Targeted chemotherapy prior to surgery; Radiation: Milestone 3: Chemoradiotherapy (cXRT); Drug: Milestone 4: standard FOLFIRINOX chemotherapy prior to surgery; Radiation: Milestone 4: Chemoradiotherapy (cXRT); Drug: Milestone 5: Targeted chemotherapy after surgery; Radiation: Milestone 5: Chemoradiotherapy (cXRT); Drug: Milestone 6: Gemcitabine after surgery; Radiation: Milestone 6: Chemoradiotherapy (cXRT); Radiation: Milestone 7: Chemoradiotherapy (cXRT); Drug: Milestone 8: Targeted chemotherapy after surgery; Drug: Milestone 9: Gemcitabine after surgery; Other: Milestone 10: No additional therapy after surgery

INTERVENTIONS:
Drug: Milestone 1: Targeted chemotherapy prior to surgery — The molecular profile from the biopsy before surgery will point to a particular chemotherapy treatment.
  Other Names: FOLFIRINOX; FOLFIRI; Gemcitabine with irinotecan; Gemcitabine / oxaliplatin; Gemcitabine / cisplatinum; Gemcitabine / capecitabine; Gemcitabine / nab-paclitaxel; Capecitabine / nab-paclitaxel
Radiation: Milestone 2: Chemoradiotherapy (cXRT) — A radio-sensitizing chemotherapy agent (either Gemcitabine or Capecitabine) will be given. Using 3D conformal or intensity-modulated radiation therapy (IMRT) techniques, patients will receive a total dose of 50.4 Gy prescribed to the 95% isodose at 1.8 Gy/fraction (28 fractions).
  Other Names: Gemcitabine; Capecitabine
Drug: Milestone 3: Targeted chemotherapy prior to surgery — The molecular profile from the biopsy before surgery will point to a particular chemotherapy treatment.
  Other Names: FOLFIRINOX; FOLFIRI; Gemcitabine with irinotecan; Gemcitabine / oxaliplatin; Gemcitabine / cisplatinum; Gemcitabine / capecitabine; Gemcitabine / nab-paclitaxel; Capecitabine / nab-paclitaxel
Radiation: Milestone 3: Chemoradiotherapy (cXRT) — A radio-sensitizing chemotherapy agent (either Gemcitabine or Capecitabine) will be given. Using 3D conformal or IMRT techniques, patients will receive a total dose of 50.4 Gy prescribed to the 95% isodose at 1.8 Gy/fraction (28 fractions).
  Other Names: Gemcitabine; Capecitabine
Drug: Milestone 4: standard FOLFIRINOX chemotherapy prior to surgery — A biopsy of the borderline tumor does not provide a molecular profile that can be used to target treatment. The treatment will be standard FOLFIRINOX chemotherapy regimen.
  Other Names: FOLFIRINOX; oxaliplatin; irinotecan; leucovorin; 5 fluorouracil
Radiation: Milestone 4: Chemoradiotherapy (cXRT) — A radio-sensitizing chemotherapy agent (either Gemcitabine or Capecitabine) will be given. Using 3D conformal or IMRT techniques, patients will receive a total dose of 50.4 Gy prescribed to the 95% isodose at 1.8 Gy/fraction (28 fractions).
  Other Names: Gemcitabine; Capecitabine
Drug: Milestone 5: Targeted chemotherapy after surgery — The molecular profile from the surgical specimen will point to a particular chemotherapy treatment.
  Other Names: FOLFIRINOX; FOLFIRI; Gemcitabine with irinotecan; Gemcitabine / oxaliplatin; Gemcitabine / cisplatinum; Gemcitabine / capecitabine; Gemcitabine / nab-paclitaxel; Capecitabine / nab-paclitaxel; Gemcitabine; Capecitabine; 5-Fluorouracil
Radiation: Milestone 5: Chemoradiotherapy (cXRT) — A radio-sensitizing chemotherapy agent (either Gemcitabine or Capecitabine) will be given. Using 3D conformal or IMRT techniques, patients will receive a total dose of 50.4 Gy prescribed to the 95% isodose at 1.8 Gy/fraction (28 fractions).
  Other Names: Gemcitabine; Capecitabine
Drug: Milestone 6: Gemcitabine after surgery — Chemotherapy treatment with Gemcitabine.
  Other Names: Chemotherapy treatment with Gemcitabine.; Gemzar
Radiation: Milestone 6: Chemoradiotherapy (cXRT) — A radio-sensitizing chemotherapy agent (either Gemcitabine or Capecitabine) will be given. Using 3D conformal or IMRT techniques, patients will receive a total dose of 50.4 Gy prescribed to the 95% isodose at 1.8 Gy/fraction (28 fractions).
  Other Names: Gemcitabine; Capecitabine
Radiation: Milestone 7: Chemoradiotherapy (cXRT) — A radio-sensitizing chemotherapy agent (either Gemcitabine or Capecitabine) will be given. Using 3D conformal or IMRT techniques, patients will receive a total dose of 50.4 Gy prescribed to the 95% isodose at 1.8 Gy/fraction (28 fractions).
  Other Names: Gemcitabine; Capecitabine
Drug: Milestone 8: Targeted chemotherapy after surgery — The molecular profile from the surgical specimen will point to a particular chemotherapy treatment.
  Other Names: FOLFIRINOX; FOLFIRI; Gemcitabine with irinotecan; Gemcitabine / oxaliplatin; Gemcitabine / cisplatinum; Gemcitabine / capecitabine; Gemcitabine / nab-paclitaxel; Capecitabine / nab-paclitaxel; Gemcitabine; Capecitabine; 5 fluorouracil
Drug: Milestone 9: Gemcitabine after surgery — Chemotherapy treatment with Gemcitabine.
  Other Names: Gemzar
Other: Milestone 10: No additional therapy after surgery — The molecular profile of the tumor that was removed during surgery points to a lack of treatment affect for available therapies. No additional therapy is recommended.
  Other Names: Restaged after surgery. No additional therapy.

SUMMARY:
In this clinical trial, if the doctor knows or suspects that a growth in the pancreas is cancer (adenocarcinoma), then a sample of the growth is tested (the test is called molecular profiling). The results of the test are used by the doctor to recommend therapy (chemotherapy and radiation therapy) that the patient will receive before having surgery to remove the adenocarcinoma. When the patient goes to surgery, the adenocarcinoma that is removed is tested again. The results of that test are used to guide the choice of therapy after surgery.

The chemotherapy drugs and the radiation therapy used in this clinical trial are already approved for treatment of pancreas cancer. This trial is intended to establish which treatment is best for a specific patient, based on test results from that patient's actual adenocarcinoma. In the past, the decision as to which treatment the patient will receive was not based on testing of the actual adenocarcinoma.

See treatment pathways at http://www.mcw.edu/surgery/patientinfo/Pancreatic-Cancer-Trial.htm.

Hypothesis: Resectability rate, overall survival rate and progression-free survival in subjects with adenocarcinoma of the pancreas will be superior for who receive targeted "personalized" therapy.

ELIGIBILITY:
Inclusion criteria:

* 18 years of age or older
* Able to understand and provide written informed consent
* Diagnosis of adenocarcinoma of the pancreas or high suspicion of adenocarcinoma of the pancreas based on CT and MRI findings as detailed below by "Definition of...."

Treatment Eligibility Criteria:

* Have an Eastern Cooperative Oncology Group performance status less than or equal to 2
* Have biopsy-proven resectable or borderline resectable adenocarcinoma of the pancreas
* Have adequate organ and bone marrow function as defined by:

  * total leukocytes greater than or equal to 3 x1000/μL
  * absolute neutrophil count (ANC) > or equal to 1.5x 1000/μL
  * hemoglobin > or equal to 9 g/dL
  * platelets > or equal to 100 x 1000/μL
  * creatinine clearance >60 mL/min or creatinine < or equal to 1.5 mg/dL
  * bilirubin < or equal to 2 mg/dL or >2 and declining as described in the protocol
  * aspartate transaminases (AST/SGOT) < or equal to3 x upper limit of normal (ULN)
  * alanine transaminases (ALT/SGPT) < or equal to 3 x ULN
* Female patients must be post menopausal for > 1 year, surgically sterile, or have a negative pregnancy test and used at least one form of contraception for 4 weeks prior to Day 1 of the study, during study treatment and during the first 4 months after study treatment is discontinued. Male patients must be surgically sterile or use barrier contraception during the study and for 4 months after the last dose of any study drug.

Definition of Resectable Pancreatic Cancer includes:

* No evidence of extra-pancreatic disease
* No evidence of tumor-arterial abutment (celiac, superior mesenteric artery or hepatic artery)
* If tumor induced narrowing of the superior mesenteric vein, portal vein or superior mesenteric-portal vein confluence is present it must be <50% of the diameter of the vessel
* Ca19-9 <5000, when bilirubin is <2 (or >2 and declining as described in the protocol)

Definition of Borderline Resectable Pancreatic Cancer to include at least one of the following:

* Tumor abutment < or equal to 180 degrees of the superior mesenteric artery or celiac axis
* Tumor abutment or encasement (>180 degrees) of a short segment of the hepatic artery
* Tumor induced narrowing of superior mesenteric vein, portal vein or superior mesenteric-portal vein of >50% of the diameter of the vessel.
* Short segment occlusion of the superior mesenteric vein, portal vein or superior mesenteric-portal vein confluence with a suitable portal vein above and superior mesenteric vein below, for reconstruction
* CT or MRI findings suspicious for, but not diagnostic of, metastatic disease (based on multidisciplinary assessment at the Medical College of Wisconsin weekly pancreatic cancer conference)
* Biopsy proven N1 disease (regional lymph nodes involved) from pre-referral biopsy or endoscopic ultrasound-guided fine needle aspirate
* Resectable tumor and cancer antigen 19-9 (CA19-9) >5000

Exclusion Criteria:

Any patient with one or more of the following will be excluded:

* Have received chemotherapy or chemoradiation within 5 years prior of study enrollment
* Have any previous history of another malignancy (other than cured basal or squamous cell carcinoma of the skin or cured in-situ carcinoma of the cervix) within 5 years of study enrollment
* Uncontrolled comorbidities including, but not limited to, ongoing or active serious infection, symptomatic congestive heart failure, unstable angina, unstable cardiac arrhythmias, psychiatric illness, excessive obesity, or situations that would limit compliance with the study requirements or the ability to willingly give written informed consent
* Known human immunodeficiency virus, hepatitis B virus, or hepatitis C virus infection
* Pregnant or breast-feeding patients or any patient with child-bearing potential not using contraception 4 weeks prior to, during and 4 months after study treatment is discontinued

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2011-11; Primary Completion 2018-06 (Actual); Study Completion 2022-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas B. Evans, M.D., FACS, Principal Investigator — Medical College of Wisconsin; Kathleen Christians, M.D., FACS, Principal Investigator — Medical College of Wisconsin; Susan Tsai, M.D., M.H.S., Principal Investigator — Medical College of Wisconsin; Paul Ritch, M.D., Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edge SB, Compton CC. The American Joint Committee on Cancer: the 7th edition of the AJCC cancer staging manual and the future of TNM. Ann Surg Oncol. 2010 Jun;17(6):1471-4. doi: 10.1245/s10434-010-0985-4. PMID 20180029
- [Result] Tsai S, Christians KK, George B, Ritch PS, Dua K, Khan A, Mackinnon AC, Tolat P, Ahmad SA, Hall WA, Erickson BA, Evans DB. A Phase II Clinical Trial of Molecular Profiled Neoadjuvant Therapy for Localized Pancreatic Ductal Adenocarcinoma. Ann Surg. 2018 Oct;268(4):610-619. doi: 10.1097/SLA.0000000000002957. PMID 30080723

RESULTS

PARTICIPANT FLOW:
Groups:
- Milestones Related to Standard Therapy: The milestones described below represent the treatment progression patients follow for treatment of this disease. The milestone represents changes in therapy based on medical condition and are not intended to represent discrete events in the investigation. Study are not parsed for analysis among the treatment milestones.
  Milestone 1: Targeted chemotherapy prior to surgery: 8 weeks targeted chemotherapy; restaging.
  Milestone 2: Before surgery: Chemoradiotherapy (cRXT); restaging Milestone 3: Before surgery: 8 weeks targeted chemotherapy; restaging; chemoradiotherapy (cXRT); restaging.
  Milestone 4: standard FOLFIRINOX chemotherapy prior to surgery: 8 weeks FOLFIRINOX (standard chemotherapy); restaging; standard chemoradiotherapy (cXRT); restaging.
  Milestone 5: After surgery: 8 weeks targeted chemotherapy; restaging; chemoradiotherapy (cXRT); restaging.
  Milestone 6: Gemcitabine after surgery: 8 weeks standard Gemcitabine (chemotherapy); restaging; chemoradiotherapy (cXRT); restaging.
  Milestone 7: After surgery: chemoradiotherapy (cXRT); restaging. Milestone 8: Gemcitabine after surgery: 8 weeks Gemcitabine (chemotherapy); restaging; 8 weeks Gemcitabine (chemotherapy); restaging.
  Milestone 9: No additional therapy after surgery. Milestone 10: After surgery no additional treatment.
Period: Overall Study
Arm/Group | Milestones Related to Standard Therapy
Started | 229
Treated | 130
Completed | 45
Not Completed | 184
Not completed — Physician Decision | 99
Not completed — Death | 85

BASELINE CHARACTERISTICS:
Arm/Group | Milestones Related to Therapy
Number analyzed (Participants) | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 58
  >=65 years | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 124
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 122
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 130

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Completing Therapy Including Surgical Resection.
Description: This outcome measure is the number of subjects completing therapy up to and including surgical resection. In this context, surgical excision of residual tumor is an option in the progression of usual care. Surgery was contraindicated for some participants. This measure is the number of subject who were eligible for and completed the surgical procedure.
Time Frame: At time of surgery (approximately 10 to 20 weeks after screening)
Measure: Count of Participants; unit: Participants
Groups:
- Milestones Related to Usual Therapy: Milestone 1: Targeted chemotherapy prior to surgery: 8 weeks targeted chemotherapy; restaging.
  Milestone 2: Before surgery: Chemoradiotherapy (cRXT); restaging Milestone 3: Before surgery: 8 weeks targeted chemotherapy; restaging; chemoradiotherapy (cXRT); restaging.
  Milestone 4: standard FOLFIRINOX chemotherapy prior to surgery: 8 weeks FOLFIRINOX (standard chemotherapy); restaging; standard chemoradiotherapy (cXRT); restaging.
  Milestone 5: After surgery: 8 weeks targeted chemotherapy; restaging; chemoradiotherapy (cXRT); restaging.
  Milestone 6: Gemcitabine after surgery: 8 weeks standard Gemcitabine (chemotherapy); restaging; chemoradiotherapy (cXRT); restaging.
  Milestone 7: After surgery: chemoradiotherapy (cXRT); restaging. Milestone 8: Gemcitabine after surgery: 8 weeks Gemcitabine (chemotherapy); restaging; 8 weeks Gemcitabine (chemotherapy); restaging.
  Milestone 9: No additional therapy after surgery. Milestone 10: After surgery no additional treatment.
Arm/Group | Milestones Related to Usual Therapy
Number analyzed (Participants) | 130
Participants | 107

2. Secondary Outcome: Overall Survival in Months
Description: This measure is the median time of survival (in months) at five years from the initiation of therapy. Results will be presented for two cohorts: subjects completing neoadjuvant therapy and surgical resection; and subjects completing neoadjuvant therapy but without surgical resection.
Time Frame: 5 years
Population: Results will be presented for two cohorts: subjects completing neoadjuvant therapy and surgical resection; and subjects completing neoadjuvant therapy but without surgical resection.
Measure: Median (Full Range); unit: Months
Groups:
- Milestones Related to Therapy (Resected): This population includes the participants who were eligible for and completed surgical resection of residual tumor. Milestone 1: Targeted chemotherapy prior to surgery: 8 weeks targeted chemotherapy; restaging.
  Milestone 2: Before surgery: Chemoradiotherapy (cRXT); restaging Milestone 3: Before surgery: 8 weeks targeted chemotherapy; restaging; chemoradiotherapy (cXRT); restaging.
  Milestone 4: standard FOLFIRINOX chemotherapy prior to surgery: 8 weeks FOLFIRINOX (standard chemotherapy); restaging; standard chemoradiotherapy (cXRT); restaging.
  Milestone 5: After surgery: 8 weeks targeted chemotherapy; restaging; chemoradiotherapy (cXRT); restaging.
  Milestone 6: Gemcitabine after surgery: 8 weeks standard Gemcitabine (chemotherapy); restaging; chemoradiotherapy (cXRT); restaging.
  Milestone 7: After surgery: chemoradiotherapy (cXRT); restaging. Milestone 8: Gemcitabine after surgery: 8 weeks Gemcitabine (chemotherapy); restaging; 8 weeks Gemcitabine (chemotherapy); restaging.
  Milestone 9: No additional therapy after surgery. Milestone 10: After surgery no additional treatment.
- Milestones Related to Therapy (Non-Resected): This population includes participants for whom surgical resection was contraindicated and did not occur.
  Milestone 1: Targeted chemotherapy prior to surgery: 8 weeks targeted chemotherapy; restaging.
  Milestone 2: Before surgery: Chemoradiotherapy (cRXT); restaging Milestone 3: Before surgery: 8 weeks targeted chemotherapy; restaging; chemoradiotherapy (cXRT); restaging.
  Milestone 4: standard FOLFIRINOX chemotherapy prior to surgery: 8 weeks FOLFIRINOX (standard chemotherapy); restaging; standard chemoradiotherapy (cXRT); restaging.
Arm/Group | Milestones Related to Therapy (Resected) | Milestones Related to Therapy (Non-Resected)
Number analyzed (Participants) | 107 | 23
Months | 45 [24 to 60] | 11 [8 to 20]

3. Secondary Outcome: Progression-free Survival
Description: This measure is the number of subjects not experiencing tumor progression at five years from initiating therapy.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Milestones Related to Usual Therapy
Number analyzed (Participants) | 130
Participants | 36

4. Secondary Outcome: Use of Biomarkers to Determine Course of Treatment
Description: The number of subjects for whom a biomarker (i.e., molecular profile) was used to determine the course of treatment.
Time Frame: Initiation of therapy (approximately 4 to 12 weeks after screening) until surgery (approximately 10 to 20 weeks after screening)
Measure: Count of Participants; unit: Participants
Arm/Group | Milestones Related to Usual Therapy
Number analyzed (Participants) | 130
Participants | 92

5. Secondary Outcome: Histologic Response to Targeted Chemotherapeutic Regimens in Resected Tumors.
Description: The number of tumors showing a histologic response. Histological response will be measured using the Ryan Score method as defined by the American Joint Committee on Cancer, 7th edition (see Edge, 2010). Grading categories are defined as: Grade 0 (complete response); Grade 1 (near complete response); Grade 2 (partial response); and Grade 3 (poor or no response).
Time Frame: At time of surgery (approximately 10 to 20 weeks after screening)
Population: Pathology results were not reported for two subject.
Measure: Count of Participants; unit: Participants
Arm/Group | Milestones Related to Usual Therapy
Number analyzed (Participants) | 107
Participants
  Complete Response | 2
  Near Complete Response | 17
  Partial Response | 44
  Poor or No Response | 42
  Results Not Available | 2

ADVERSE EVENTS:
Time Frame: 5 years
Description: The treatment milestones are represent the usual care for this condition. Only serious adverse events were collected.
Arm/Group | Milestones Related to Therapy
All-Cause Mortality (participants affected / at risk) | 85/130
Serious Adverse Events (participants affected / at risk) | 50/130
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milestones Related to Therapy (N=130)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Febrile neutorpenia (Blood and lymphatic system disorders) | 3 (3)
Acute coronary syndrome (Cardiac disorders) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 3 (3)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Duodenal obstruction (Gastrointestinal disorders) | 2 (2)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1)
Jejunal obstruction (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Fever (General disorders) | 3 (3)
Flu-like symptoms (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 3 (3)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 3 (3)
Biliary tract infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 12 (12)
Skin infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Hyperglycemia (Investigations) | 1 (1)
Hyponatremia (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Suicidal attempt (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 4 (4)
Thromboembolic event (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT01726582/Prot_SAP_000.pdf
  • Informed Consent Form (2017-02-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT01726582/ICF_001.pdf